CLINICAL TRIAL: NCT02096575
Title: Nitrous Oxide for Pain Management of First Trimester Surgical Abortion
Acronym: NAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Rameet Singh, Assistant Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: UNMHSC12-313
Record Dates: First submitted 2014-03-20; First posted 2014-03-26 (Estimated); Results first posted 2016-03-11 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Abortion in First Trimester
Keywords: nitrous oxide; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitrous oxide administration (Experimental): All participants will receive 800 mg of oral ibuprofen 30 minutes pre-operatively. All patients will receive local anesthesia via a standardized paracervical block with 18 cc of 1% lidocaine buffered with 2 ml of 8.4% sodium bicarbonate and 0.2 ml of 4 units of vasopressin.
  In addition, the Nitrous oxide group will receive two placebo pills. Nitrous oxide will be administered via a disposable scented nasal mask to blind patients to the intervention. Nitrous oxide will be administered at a fixed ratio of 60% nitrous oxide and 40% oxygen. The nasal mask will be placed on the patient's nose and the nitrous oxide will be administered continuously.
  Interventions: Other: Nitrous oxide administration
- Standard care group (No Intervention): All participants will receive 800 mg of oral ibuprofen 30 minutes pre-operatively. All patients will receive local anesthesia via a standardized paracervical block with 18 cc of 1% lidocaine buffered with 2 ml of 8.4% sodium bicarbonate and 0.2 ml of 4 units of vasopressin.
  The standard care group will receive one 5/325 mg Percocet, and 1 mg of lorazepam, 30 minutes before the procedure. The standard care group will receive oxygen by mask intraoperatively.

INTERVENTIONS:
Other: Nitrous oxide administration — All participants will receive 800 mg of oral ibuprofen 30 minutes pre-operatively. The NO group will get two placebo pills and the standard care group will get one 5/325 mg Vicodin, and 1 mg of Ativan 30 minutes before the procedure. The standard care group will get oxygen intraoperatively.
  NO or oxygen will be administered via a scented nasal mask to blind patients to the intervention.
  All patients will get local anesthesia via a standardized PCB.
  Arms: Nitrous oxide administration

SUMMARY:
The purpose of this research is to study the effect of nitrous oxide on pain felt by women having a surgical termination at less than 11 weeks compared to pain felt by women receiving oral pain medications.

DETAILED DESCRIPTION:
This study has important implications in the field of pain management for surgical abortion. While NO is administered in some outpatient clinics for surgical abortion, its effect on pain has not been systematically studied in a randomized controlled trial in women undergoing first trimester surgical abortion under local/oral analgesia. Expanding pain management options for women undergoing abortion confers significant public health benefits.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older,
* elective pregnancy termination at gestational age of less than 11 weeks,
* speak English
* candidate for an in-clinic procedure.
* desire local anesthesia, ibuprofen, Vicodin and Ativan (the usual treatment in our clinic) for managing pain

Exclusion Criteria:

* no medical problems preventing the use of nitrous oxide
* no allergies to nitrous oxide, lidocaine, vasopressin, ibuprofen, Vicodin or Ativan
* significant active upper respiratory infection
* chronic obstructive pulmonary disease (COPD)
* intoxication
* use of street drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rameet H. Singh, MD, MPH, Principal Investigator — University of New Mexico Health Sciences Center
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Singh RH, Espey E, Carr S, Pereda B, Ogburn T, Leeman L. Nitrous oxide for pain management of first trimester surgical abortion -- a randomized controlled pilot study. Contraception. 2015 Feb;91(2):164-6. doi: 10.1016/j.contraception.2014.09.013. Epub 2014 Oct 22. PMID 25459096

RESULTS

PARTICIPANT FLOW:
Groups:
- Nitrous Oxide Administration: All participants will receive 800 mg of oral ibuprofen 30 minutes pre-operatively. All patients will receive local anesthesia via a standardized paracervical block with 18 cc of 1% lidocaine buffered with 2 ml of 8.4% sodium bicarbonate and 0.2 ml of 4 units of vasopressin.
  In addition, the Nitrous oxide group will receive two placebo pills. Nitrous oxide will be administered via a disposable scented nasal mask to blind patients to the intervention. Nitrous oxide will be administered at a fixed ratio of 60% nitrous oxide and 40% oxygen. The nasal mask will be placed on the patient's nose and the nitrous oxide will be administered continuously.
  Nitrous oxide administration
- Excluded: Participants that were withdrawn from the study after consent
Period: Overall Study
Arm/Group | Nitrous Oxide Administration | Standard Care Group | Excluded
Started | 68 | 67 | 5
Completed | 68 | 67 | 0
Not Completed | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitrous Oxide Administration | Standard Care Group | Total
Number analyzed (Participants) | 68 | 67 | 135
Age, Customized [Mean (Full Range); unit: years] | 26.72 [18 to 48] | 26.03 [18 to 42] | 26.38 [18 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 67 | 135
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 3 | 3
  Black or African American | 2 | 3 | 5
  Native American/ Alaska Native | 12 | 4 | 16
  Native Hawaiian/ Pacific Islander | 1 | 0 | 1
  Hispanic/ Latino | 9 | 5 | 14
  White | 37 | 45 | 82
  Bi or Multiracial | 5 | 4 | 9
  Other | 1 | 0 | 1
  Unknown or Not reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 68 | 67 | 135

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Pain Score for Mean Maximum Procedural Pain
Description: The primary outcome of this study is to evaluate the difference in mean maximum pain experienced during the procedure between groups as assessed 5 minutes after the procedure is completed.
  Pain was assessed using the Visual Analog Scale (VAS). 0 = no pain, 100 = maximum pain
Time Frame: Mean maximum pain experienced during the procedure and assessed 5 minutes after the procedure
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Nitrous Oxide Administration | Standard Care Group
Number analyzed (Participants) | 68 | 67
units on a scale | 54.37 [3 to 100] | 60.48 [1 to 100]

2. Secondary Outcome: Visual Analog Scale Score for Baseline Pain
Description: A quantitative assessment of pain prior to the procedure. Pain was assessed using the Visual Analog Scale (VAS). 0 = no pain, 100 = maximum pain
Time Frame: Baseline pain assessment on average within 30 minutes before procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Nitrous Oxide Administration: All participants will receive 800 mg of oral ibuprofen 30 minutes pre-operatively. All patients will receive local anesthesia via a standardized paracervical block with 18 cc of 1% lidocaine buffered with 2 ml of 8.4% sodium bicarbonate and 0.2 ml of 4 units of vasopressin.
  The Nitrous oxide group will receive two placebo pills. Nitrous oxide will be administered via a disposable scented nasal mask to blind patients to the intervention. Nitrous oxide will be administered at a fixed ratio of 60% nitrous oxide and 40% oxygen. The nasal mask will be placed on the patient's nose and the nitrous oxide will be administered continuously.
  Nitrous oxide administration: The NO group will get two placebo pills.
Arm/Group | Nitrous Oxide Administration | Standard Care Group
Number analyzed (Participants) | 68 | 67
units on a scale | 4.7426 (12.884) | 4.4388 (11.7748)

3. Secondary Outcome: Visual Analog Scale for Post-procedure Pain
Description: A quantitative assessment of post-procedure pain. Pain was assessed using the Visual Analog Scale (VAS). 0 = no pain, 100 = maximum pain
Time Frame: Visual analog scale administered on average 20 minutes after procedure completed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nitrous Oxide Administration | Standard Care Group
Number analyzed (Participants) | 68 | 67
units on a scale | 26.68 (22.28) | 25.96 (24.33)

4. Secondary Outcome: Pain Management Satisfaction
Description: Quantitative assessment of pain management. Pain was assessed using the Visual Analog Scale (VAS). 0 = no pain, 100 = maximum pain
Time Frame: Visual analog scale for satisfaction administered on average within 20 minutes after procedure completion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nitrous Oxide Administration | Standard Care Group
Number analyzed (Participants) | 68 | 67
units on a scale | 69.3382 (28.3789) | 61.5373 (30.3536)

5. Secondary Outcome: Visual Analog Scale to Measure Anticipated Pain.
Description: Anticipated pain is assessed before the procedure. Pain was assessed using the Visual Analog Scale (VAS). 0 = no pain, 100 = maximum pain
Time Frame: Anticipated pain assessed on average within 30 minutes before procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nitrous Oxide Administration | Standard Care Group
Number analyzed (Participants) | 68 | 67
units on a scale | 56.1544 (24.4817) | 50.3104 (21.7043)

ADVERSE EVENTS:
Arm/Group | Nitrous Oxide Administration | Standard Care Group
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/67
Other Adverse Events (participants affected / at risk) | 0/68 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No